CLINICAL TRIAL: NCT01491035
Title: An Open-label Study Evaluating the Pharmacokinetics and Tolerability of [Vortioxetine] Lu AA21004 in Connection With Multiple Oral Dosing of [Vortioxetine] Lu AA21004 in Child and Adolescent Patients With a DSM-IV Diagnosis of Depressive or Anxiety Disorder
Brief Title: Pharmacokinetics and Tolerability of Vortioxetine (Lu AA21004) in Child and Adolescent Patients With Depressive or Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12708A; 2010-020170-42 (EudraCT Number)
Record Dates: First submitted 2011-11-23; First posted 2011-12-13 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Depressive Disorder; Anxiety Disorder
Keywords: Children; Adolescents; Pharmacokinetic; Pharmacodynamic
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort CC1, 6 children (Experimental)
  Interventions: Drug: Vortioxetine
- Cohort CC2, 6 children (Experimental)
  Interventions: Drug: Vortioxetine
- Cohort CC3, 6 children (Experimental)
  Interventions: Drug: Vortioxetine
- Cohort CC4, 6 children (Experimental)
  Interventions: Drug: Vortioxetine
- Cohort AC1, 6 adolescents (Experimental)
  Interventions: Drug: Vortioxetine
- Cohort AC2, 6 adolescents (Experimental)
  Interventions: Drug: Vortioxetine
- Cohort AC3, 6 adolescents (Experimental)
  Interventions: Drug: Vortioxetine
- Cohort AC4, 6 adolescents (Experimental)
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — 5 mg tablets for 14 days; orally; once daily
  Other Names: Brintellix
  Arms: Cohort AC1, 6 adolescents; Cohort CC1, 6 children
Drug: Vortioxetine — 10 mg tablets for 14 days (initial up-titration with 5 mg/day for 2 days); orally; once daily
  Other Names: Brintellix
  Arms: Cohort AC2, 6 adolescents; Cohort CC2, 6 children
Drug: Vortioxetine — 15 mg tablets for 14 days (initial up-titration with 5 and 10 mg/day for a total of 4 days); orally; once daily
  Other Names: Brintellix
  Arms: Cohort AC3, 6 adolescents; Cohort CC3, 6 children
Drug: Vortioxetine — 20 mg tablets for 14 days (initial up-titration with 5, 10, and 15 mg/day for a total of 6 days); orally; once daily
  Other Names: Brintellix
  Arms: Cohort AC4, 6 adolescents; Cohort CC4, 6 children

SUMMARY:
The objective of the study is to evaluate the pharmacokinetics of vortioxetine and its metabolites in connection with multiple oral dosing in child and adolescent patients with a DSM-IV-TR diagnosis of Depressive or Anxiety Disorder

DETAILED DESCRIPTION:
The study will be conducted in the US and in Europe and will include paediatric patients diagnosed with depressive or anxiety disorders of two age populations; children aged 7-11 years and adolescents of the age 12-17 years. It is an open study to allow pharmacokinetic (PK) sampling of all patients and four dose levels will be tested. Following lower initial doses for 2 to 6 days, the patients will be treated once daily at the assigned dose levels for 14 days, and it is expected that patients may benefit from treatment during this period. As the treatment duration is not sufficient according to treatment guidelines, if judged or indicated by the investigator, the patients are offered to continue in an extension treatment of up to six months to allow possibility for therapeutic satisfaction.

Preferably, the cohorts will be dosed in the following order: AC1, AC2, CC1, AC3, CC2, AC4, CC3, and CC4. An external data safety monitoring board (DSMB) will be established to evaluate safety, tolerability and preliminary PK data from the dosed cohort(s) prior to any dosing of subsequent cohort (s). The dose regimen may be adjusted based on the recommendation of the DSMB. Adolescents will be exposed to a certain dose of vortioxetine before children receive the same dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a DSM-IV-TR diagnosis of Depressive or Anxiety Disorder.
* The patient and parent(s)/legal representative(s) are able to comprehend and satisfactorily comply with the protocol requirements.
* Treatment with antidepressant therapy is warranted, as judged by the investigator.

Exclusion Criteria:

* The patient is pregnant or breast-feeding.
* The patient presents or has a history of an Axis I (DSM-IV-TR) diagnosis of Bipolar Disorder, Post Traumatic Stress Disorder (PTSD), Autism, Pervasive Developmental Disorder (PDD), Obsessive Compulsive Disorder (OCD) or Schizophrenia or Schizoaffective Disorder.
* The patient has not maintained a stable dose of a methylphenidate or amphetamine for their treatment of attention-deficit/hyperactivity disorder (ADHD) for a minimum of 4 weeks prior to the study treatment.
* The patient has a known mental retardation, or clinical evidence or known social or school history indicative of mental retardation.
* The patient is at significant risk of committing suicide based on history (for example previous suicide attempt) or according to the investigator's experience, or based on active suicidal ideation, intent or plan, item 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS).
* The subject has any concurrent illness that may affect the particular target or absorption, distribution, and elimination of the investigational medicinal product (IMP).
* The patient meets DSM-IV-TR criteria for any psychoactive substance or alcohol use disorder.

Other inclusion and exclusion criteria may apply.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (7):
- United States (4):
  - US003, Washington D.C., District of Columbia
  - US004, Wichita, Kansas
  - US002, Cincinnatti, Ohio
  - US001, Cleveland, Ohio
- Germany (3):
  - DE002, Berlin
  - DE001, Mainz
  - DE003, Ulm

REFERENCES:
- [Derived] Findling RL, Robb AS, DelBello MP, Huss M, McNamara NK, Sarkis EH, Scheffer RE, Poulsen LH, Chen G, Lemming OM, Auby P. A 6-Month Open-Label Extension Study of Vortioxetine in Pediatric Patients with Depressive or Anxiety Disorders. J Child Adolesc Psychopharmacol. 2018 Feb;28(1):47-54. doi: 10.1089/cap.2017.0047. Epub 2017 Oct 16. PMID 29035574
- See also: EMA EudraCT Results: 2010-020170-42 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2010-020170-42/results

RESULTS

PARTICIPANT FLOW:
Groups:
- Adolescents, 5 mg; Children, 5 mg: Vortioxetine: 5 mg tablets for 14 days; orally; once daily
- Adolescents, 10 mg; Children, 10 mg: Vortioxetine: 10 mg tablets for 14 days (initial up-titration with 5 mg/day for 2 days); orally; once daily
- Adolescents, 15 mg; Children, 15 mg: Vortioxetine: 15 mg tablets for 14 days (initial up-titration with 5 and 10 mg/day for a total of 4 days); orally; once daily
- Adolescents, 20 mg; Children, 20 mg: Vortioxetine: 20 mg tablets for 14 days (initial up-titration with 5, 10, and 15 mg/day for a total of 6 days); orally; once daily
Period: Overall Study
Arm/Group | Adolescents, 5 mg | Adolescents, 10 mg | Adolescents, 15 mg | Adolescents, 20 mg | Children, 5 mg | Children, 10 mg | Children, 15 mg | Children, 20 mg
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adolescents, 5 mg | Adolescents, 10 mg | Adolescents, 15 mg | Adolescents, 20 mg | Children, 5 mg | Children, 10 mg | Children, 15 mg | Children, 20 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.9) | 15.3 (1.9) | 15.2 (1.2) | 14.8 (1.9) | 10.3 (1.2) | 9.7 (1.2) | 10.5 (0.8) | 9.8 (1.8) | 12.7 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 4 | 3 | 3 | 2 | 2 | 25
  Male | 3 | 3 | 1 | 2 | 3 | 3 | 4 | 4 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 1 | 4 | 3 | 2 | 16
  White | 4 | 4 | 4 | 4 | 4 | 2 | 3 | 4 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 3 | 4 | 6 | 6 | 6 | 43
  Germany | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Vortioxetine
Description: Maximum plasma concentration of vortioxetine
Time Frame: Pre-dose and 1, 3, 5, 8, 12 and 24 hours post-dose on Day 14, 16, 18, or 20, depending on assigned dose level
Population: Pharmacokinetic analysis set = all patients who took at least one dose of IMP and who contributed with both Day 1 pre-dose pharmacokinetic sampling data and sufficient post-dose sampling data for estimation of the pharmacokinetic parameters.
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Adolescents, 5 mg | Adolescents, 10 mg | Adolescents, 15 mg | Adolescents, 20 mg | Children, 5 mg | Children, 10 mg | Children, 15 mg | Children, 20 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 4.3 (3.7) | 7.8 (2.8) | 15 (6.2) | 16 (8.1) | 5.0 (3.3) | 14 (8.2) | 26 (21) | 31 (20)

2. Primary Outcome: AUC(0-24h) of Vortioxetine
Description: Area under the vortioxetine plasma concentration-time curve from 0 to 24 hours
Time Frame: Pre-dose and 1, 3, 5, 8, 12 and 24 hours post-dose on Day 14, 16, 18 or 20, depending on assigned dose level
Population: Pharmacokinetic analysis set
Measure: Median (Standard Deviation); unit: ng*h/mL
Arm/Group | Adolescents, 5 mg | Adolescents, 10 mg | Adolescents, 15 mg | Adolescents, 20 mg | Children, 5 mg | Children, 10 mg | Children, 15 mg | Children, 20 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 82 (71) | 144 (60) | 283 (115) | 304 (143) | 89 (66) | 261 (137) | 492 (373) | 562 (374)

3. Primary Outcome: t½ of Vortioxetine
Description: Half-life of vortioxetine in plasma
Time Frame: Pre-dose and 1, 3, 5, 8, 12 and 24 hours post-dose on Day 14, 16, 18 or 20, depending on assigned dose level
Population: Pharmacokinetic analysis set
Measure: Median (Standard Deviation); unit: h
Arm/Group | Adolescents, 5 mg | Adolescents, 10 mg | Adolescents, 15 mg | Adolescents, 20 mg | Children, 5 mg | Children, 10 mg | Children, 15 mg | Children, 20 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h | 46 (33) | 56 (19) | 50 (16) | 40 (10) | 45 (27) | 52 (18) | 71 (52) | 62 (23)

4. Primary Outcome: Cmax of Lu AA34443
Description: Maximum plasma concentration of the major, inactive metabolite Lu AA34443
Time Frame: Pre-dose and 1, 3, 5, 8, 12 and 24 hours post-dose on Day 14, 16, 18, or 20, depending on assigned dose level
Population: Pharmacokinetic analysis set
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Adolescents, 5 mg | Adolescents, 10 mg | Adolescents, 15 mg | Adolescents, 20 mg | Children, 5 mg | Children, 10 mg | Children, 15 mg | Children, 20 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 3.5 (2.2) | 14 (7.1) | 16 (5.3) | 38 (12) | 7.8 (3.4) | 15 (5.4) | 20 (13) | 47 (17)

5. Primary Outcome: AUC(0-24h) of Lu AA34443
Description: Area under the plasma concentration-time curve from 0 to 24 hours for the major, inactive metabolite Lu AA34443
Time Frame: Pre-dose and 1, 3, 5, 8, 12 and 24 hours post-dose on Day 14, 16, 18 or 20, depending on assigned dose level
Population: Pharmacokinetic analysis set
Measure: Median (Standard Deviation); unit: ng*h/mL
Arm/Group | Adolescents, 5 mg | Adolescents, 10 mg | Adolescents, 15 mg | Adolescents, 20 mg | Children, 5 mg | Children, 10 mg | Children, 15 mg | Children, 20 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 56 (29) | 223 (98) | 266 (100) | 544 (192) | 115 (47) | 241 (93) | 429 (232) | 646 (251)

6. Primary Outcome: t½ of Lu AA34443
Description: Half-life of the major, inactive metabolite Lu AA34443 in plasma
Time Frame: Pre-dose and 1, 3, 5, 8, 12 and 24 hours post-dose on Day 14, 16, 18 or 20, depending on assigned dose level
Population: Pharmacokinetic analysis set
Measure: Median (Standard Deviation); unit: h
Arm/Group | Adolescents, 5 mg | Adolescents, 10 mg | Adolescents, 15 mg | Adolescents, 20 mg | Children, 5 mg | Children, 10 mg | Children, 15 mg | Children, 20 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h | 26 (9.3) | 33 (13) | 24 (11) | 24 (5.1) | 20 (24) | 19 (9.6) | 29 (6.1) | 27 (8.8)

7. Primary Outcome: Oral Clearance (CL/F) of Vortioxetine
Description: Oral clearance expressed as a function of bioavailability
Time Frame: Pre-dose and 1, 3, 5, 8, 12 and 24 hours post-dose on Day 14, 16, 18 or 20, depending on assigned dose level
Population: Pharmacokinetic analysis set
Measure: Median (Standard Deviation); unit: L/h
Arm/Group | Adolescents, 5 mg | Adolescents, 10 mg | Adolescents, 15 mg | Adolescents, 20 mg | Children, 5 mg | Children, 10 mg | Children, 15 mg | Children, 20 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
L/h | 60 (55) | 50 (16) | 50 (23) | 61 (20) | 50 (16) | 42 (25) | 29 (33) | 34 (17)

ADVERSE EVENTS:
Time Frame: 4 to 5 weeks, depending on the assigned dose
Arm/Group | Adolescents, 5 mg | Adolescents, 10 mg | Adolescents, 15 mg | Adolescents, 20 mg | Children, 5 mg | Children, 10 mg | Children, 15 mg | Children, 20 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 5/6 | 5/6 | 5/6 | 5/6 | 5/6 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adolescents, 5 mg (N=6) | Adolescents, 10 mg (N=6) | Adolescents, 15 mg (N=6) | Adolescents, 20 mg (N=6) | Children, 5 mg (N=6) | Children, 10 mg (N=6) | Children, 15 mg (N=6) | Children, 20 mg (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 2 | 2 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritability (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pica (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 2 | 1 | 2 | 0 | 2 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 1 | 1 | 3 | 2 | 3 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Frustration (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hostility (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No